CLINICAL TRIAL: NCT05721807
Title: Effectiveness of Functional Magnetic Stimulation and Pelvic Floor Muscle Training on Pelvic Floor Muscle Function, Urinary Incontinence Symptoms and Quality of Life in Women With Stress Urinary Incontinence
Brief Title: Physiotherapy in Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LithuanianSportsU-13
Record Dates: First submitted 2023-01-19; First posted 2023-02-10 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Urinary Incontinence,Stress
Keywords: stress incontinence; pelvic floor; functional magnetic stimulation; muscle training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- functional magnetic stimulation (Experimental): functional magnetic stimulation for stress urinary incontinence
  Interventions: Other: functional magnetic stimulation
- pelvic floor muscle training program (Experimental): exercise program for pelvic floor muscle
  Interventions: Other: pelvic floor muscle training program

INTERVENTIONS:
Other: functional magnetic stimulation — When applying functional magnetic stimulation, the stress urinary incontinence program "P2 stress" was chosen. The first 20 min. current frequency was 35 Hz, modulation - rising amplitude (from 0 to maximum per second), total wave duration 12 s. active time 6 s., pause time 6 s. After 20 min. current frequency changed to 5 Hz, modulation and wave remained the same. After 2 min. current frequency changed to 35 Hz, modulation - amplitude, one-sided sinusoidal, wave remained the same. The total duration of the procedure was 30 min. A magnetic spring is installed at the bottom of the chair. During the treatment, each subject was instructed to sit on a chair so that the perineum was centered on the spring and that the subjects felt the contraction of the muscles. The intensity of the magnetic field was adjusted so as to feel comfortable during the study procedure (Vadalà et al., 2017).
  Arms: functional magnetic stimulation
Other: pelvic floor muscle training program — The program consisted of two parts. From procedures 1 to 6, 6 exercises were performed, after 6 times the exercises were adjusted, and from procedures 7 to 12, another 5 exercises were performed. The program consists of breathing, pelvic floor muscle strength, endurance, speed training exercises and exercises to strengthen the thighs, buttocks, deep back and deep abdominal muscles. Exercises were performed in 2 sets of 10 repetitions at an intensity from various positions: lying on the back, side, sitting, quadruped (Oliveira et al., 2017; Walton et al., 2019).
  Arms: pelvic floor muscle training program

SUMMARY:
The goal of this randomized controlled trial is to evaluate and compare the effects of functional magnetic stimulation and pelvic floor muscle training on pelvic floor muscle function, urinary incontinence symptoms and quality of life in women with stress urinary incontinence. The main questions it aims to answer are:

* What is the effect of functional magnetic stimulation on pelvic floor muscle function, symptoms of urinary incontinence and quality of life in women with stress urinary incontinence?
* What is the effect of pelvic floor muscle training program on pelvic floor muscle function, symptoms of urinary incontinence and quality of life in women with stress urinary incontinence?
* Which intervention is more effective - functional magnetic stimulation or pelvic floor muscle training program?

Participants will be evaluated before and after the intervention with the following methods:

* International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF);
* Incontinence Impact Questionnaire-Short Form (IIQ-7);
* Pelvic floor muscle strength and endurance will be assessed with a "Pelvexiser" perineometer.

DETAILED DESCRIPTION:
The study was performed in the period of 07/21/2021-30/10/2021. The study included 48 women 29-49 years old who have complained of stress urinary incontinence for at least 4 weeks, who gave birth and signed the consent form. Women complaining of vaginismus, suffering from urinary tract infection, cancer, epilepsy or skin conditions with implanted pacemakers, metal implants and pregnant women were excluded from the study. Study participants were randomly divided into two groups: the I group (n=24), in which participants underwent functional magnetic stimulation (FMS) and the II group (n=24) in which subjects received pelvic floor muscle training (PFMT) program. Participants were evaluated before the intervention and repeated after 6 weeks. Subjects responded to a general questionnaire before the intervention, before and after the intervention, the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) and Incontinence Impact Questionnaire-Short Form (IIQ-7) were used to assess the symptoms of urinary incontinence and their impact on quality of life. Pelvic floor muscle strength and endurance were assessed with a "Pelvexiser" perineometer. Statistical analysis was performed by IBM SPSS Statistics 26.0 and Microsoft Excel software 365.

ELIGIBILITY:
Inclusion Criteria:

* complains of stress incontinence for at least 4 weeks;
* women who have given birth.

Exclusion Criteria:

* pregnancy;
* vaginism;
* urinal infection;
* oncological disorders;
* epilepsy;
* skin problems;
* if they had an implanted heart pacemaker, metal implants.

Ages: 29 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence symptoms and quality of life (International Consultation on Incontinence Questionnaire) | Change from Baseline Urinary Incontinence symptoms at 6 weeks
  ICIQ - SF - International Consultation on Incontinence Questionnaire - Short Form is intended to subjectively evaluate the symptoms of urinary incontinence in a woman or man and the impact of those symptoms on the quality of life. The questionnaire consists of four questions. The first two questions assess the symptoms of urinary incontinence experienced, the third question describes quality of life and the fourth question determines which type of incontinence the person has. The scores of the first three questions are summed up, the maximum number of points collected is 21, the minimum is 0. Depending on the number of points collected, the severity of urinary incontinence symptoms is assessed: no urinary incontinence symptoms (0 points), mild urinary incontinence symptoms (1 - 5 points), moderate incontinence symptoms (score 6-12), severe incontinence symptoms (score 13-18) and very severe incontinence symptoms (19-21).
IIQ-7 -Incontinence Impact Questionnaire | Change from Baseline Incontinence Impact Questionnaire scores at 6 weeks
  The IIQ-7 questionnaire is designed to assess the impact of urinary incontinence on quality of life. The questionnaire consists of seven questions, which can be answered to find out the impact of urinary incontinence on all areas of life: physical activity, traveling, social activity, relationships, emotional state. Each question is evaluated from 0 to 3 points. The higher the score, the worse the quality of life. The maximum number of collected points is 100, the minimum is 0. <50 points is considered a good quality of life, 50-70 points is an average quality of life, >70 points is a poor quality of life.
Perineometry | Change from Baseline Perineometry at 6 weeks
  The strength and endurance of the subjects' pelvic floor muscles was assessed with a Pelvexiser perineometer (Wolfram Haboeck Co., Austria). This apparatus has been scientifically proven as an objective method of assessing the function of the pelvic floor muscles and an effective exerciser for strengthening the pelvic floor muscles, which is why it is often used in the presence of for urinary incontinence problems. The Pelvexiser can provide varying resistance to the pelvic floor muscles and provide real-time feedback on pelvic floor muscle contractions and changes (Chitra et al., 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Dudonienė, Study Chair — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No